CLINICAL TRIAL: NCT01365455
Title: A Randomized, Double-blind, Placebo Controlled, Multicenter Study of Subcutaneous Secukinumab to Demonstrate Efficacy After Twelve Weeks of Treatment, and to Assess the Safety, Tolerability and Long-term Efficacy up to One Year in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis
Brief Title: Efficacy and Safety of Subcutaneous Secukinumab for Moderate to Severe Chronic Plaque-type Psoriasis for up to 1 Year
Acronym: ERASURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457A2302; 2010-023512-13 (EudraCT Number)
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2019-03

CONDITIONS: Moderate to Severe Plaque-type Psoriasis
Keywords: Psoriasis; plaque; plaque-type psoriasis; IL-17 blocker; subcutaneous; psoriatic arthritis; injection; AIN457; AIN457A; secukinumab
MeSH Terms: conditions — Psoriasis; Plaque, Amyloid; Arthritis, Psoriatic | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- AIN457 150 mg (Experimental): AIN457 secukinumab 150 mg subcutaneous (s.c.) injection plus a placebo secukinumab s.c. injection once weekly for 4 weeks (at randomization, Weeks 1, 2, and 3), followed by dosing every 4 weeks, starting at Week 4 and until Week 48, except for Weeks 13, 14, and 15 when they received two s.c. injections of placebo per week
  Interventions: Drug: secukinumab 150 mg; Drug: placebo to secukinumab 150 mg
- AIN457 300 mg (Experimental): AIN457 secukinumab 300 mg (two s.c. injections of 150 mg) once weekly for 4 weeks (at randomization, Weeks 1, 2, and 3), followed by dosing every 4 weeks, starting at Week 4, and until Week 48, except for Weeks 13, 14, and 15 when they received two s.c. injections of placebo per week
  Interventions: Drug: secukinumab 150 mg; Drug: placebo to secukinumab 150 mg
- placebo (Placebo Comparator): placebo secukinumab (two s.c. injections per dose) once weekly for 4 weeks (at randomization, Weeks 1, 2, and 3), followed by dosing every 4 weeks (Weeks 4 and 8). Prior to receiving the Week 12 dose, all patients in the placebo group were assigned to the following treatment groups based on their PASI 75 response at Week 12. PASI 75 responders: continued on placebo and received their placebo injections at Weeks 12, 13, 14, 15, and then every 4 weeks starting at Week 16 until Week 48.
  Interventions: Drug: placebo to secukinumab 150 mg
- AIN457 150mg from Placebo (Experimental): Patients randomized to AIN457 150mg in Maintenance phase when they were on Placebo in Induction Phase because they were PASI 75 non-responders and received their treatment on Weeks 12, 13, 14, 15, and then every 4 weeks starting at Week 16 until Week 48.
  Interventions: Drug: secukinumab 150 mg; Drug: placebo to secukinumab 150 mg
- AIN457 300mg from Placebo (Experimental): Patients randomized to AIN457 300mg in Maintenance phase when they were on Placebo in Induction Phase. PASI 75 non-responders and received their treatment on Weeks 12, 13, 14, 15, and then every 4 weeks starting at Week 16 until Week 48.
  Interventions: Drug: secukinumab 150 mg; Drug: placebo to secukinumab 150 mg

INTERVENTIONS:
Drug: secukinumab 150 mg — secukinumab (AIN457) 150mg or 300mg subcutaneous
  Arms: AIN457 150 mg; AIN457 150mg from Placebo; AIN457 300 mg; AIN457 300mg from Placebo
Drug: placebo to secukinumab 150 mg — Placebo to Match secukinumab (AIN457) 150mg or 300mg subcutaneous

SUMMARY:
This study will assess the safety and efficacy of secukinumab compared to placebo in patients that have moderate to severe, chronic, plaque-type psoriasis.

ELIGIBILITY:
Inclusion criteria:

* Moderate and severe plaque-type psoriasis diagnosed for at least 6 months.
* Severity of psoriasis disease meeting all of the following three criteria:
* Psoriasis Area and Severity Index (PASI) score of 12 or greater,
* Investigator's Global Assessment (IGA) score of 3 or greater,
* Total body surface area (BSA) affected of 10% or greater.
* Inadequate control by prior use of topical treatment, phototherapy and/or systemic therapy.

Exclusion criteria:

* Current forms of psoriasis other than chronic plaque-type psoriasis (for example, pustular, erythrodermic, guttate).
* Current drug-induced psoriasis.
* Previous use of secukinumab or any drug that targets IL-17 or IL-17 receptor.
* Significant medical problems such as uncontrolled hypertension, congestive heart failure or a condition that significantly immunocompromises the subject.
* Hematological abnormalities.
* History of an ongoing, chronic or recurrent infectious disease, or evidence of untreated tuberculosis.
* History of lymphoproliferative disease or history of malignancy of any organ system within the past 5 years.
* Pregnant or nursing (lactating) women.
* Subjects not willing to limit UV light exposure during the study Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 738 (Actual)
Dates: Start 2011-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmceuticals, Study Director — Novartis Pharmaceuticals
Locations (75):
- United States (29):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Oceanside, California
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Boca Raton, Florida
  - Novartis Investigative Site, Snellville, Georgia
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Oregon City, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Bryan, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Norfolk, Virginia
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Mendoza
- Canada (5):
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Peterborough, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Colombia (4):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Bucaramanga
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Novartis Investigative Site, Kopavogur, Iceland
- Israel (3):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
- Japan (17):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Inashiki-gun, Ibaraki
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Kyoto
- Latvia (3):
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Riga
  - Novartis Investigative Site, Ventspils
- Lithuania (3):
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Vilnius
- Mexico (3):
  - Novartis Investigative Site, Zapopan, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
- Taiwan (3):
  - Novartis Investigative Site, Taoyuan District, Taiwan
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei

REFERENCES:
- [Derived] Sticherling M, Nikkels AF, Hamza AM, Kwong P, Szepietowski JC, El Sayed M, Ghislain PD, Khotko AA, Patekar M, Ortmann CE, Forrer P, Papanastasiou P, Keefe D. Secukinumab in Pediatric Patients with Plaque Psoriasis: Pooled Safety Analysis from Two Phase 3 Randomized Clinical Trials. Am J Clin Dermatol. 2023 Sep;24(5):821-835. doi: 10.1007/s40257-023-00782-8. Epub 2023 Jun 21. PMID 37341961
- [Derived] Merola JF, McInnes IB, Deodhar AA, Dey AK, Adamstein NH, Quebe-Fehling E, Aassi M, Peine M, Mehta NN. Effect of Secukinumab on Traditional Cardiovascular Risk Factors and Inflammatory Biomarkers: Post Hoc Analyses of Pooled Data Across Three Indications. Rheumatol Ther. 2022 Jun;9(3):935-955. doi: 10.1007/s40744-022-00434-z. Epub 2022 Mar 19. PMID 35305260
- [Derived] Houghton K, Patil D, Gomez B, Feldman SR. Correlation Between Change in Psoriasis Area and Severity Index and Dermatology Life Quality Index in Patients with Psoriasis: Pooled Analysis from Four Phase 3 Clinical Trials of Secukinumab. Dermatol Ther (Heidelb). 2021 Aug;11(4):1373-1384. doi: 10.1007/s13555-021-00564-2. Epub 2021 Jun 10. PMID 34110605
- [Derived] Dehlin M, Fasth AER, Reinhardt M, Jacobsson LTH. Impact of psoriasis disease activity and other risk factors on serum urate levels in patients with psoriasis and psoriatic arthritis-a post-hoc analysis of pooled data from three phase 3 trials with secukinumab. Rheumatol Adv Pract. 2021 Feb 18;5(1):rkab009. doi: 10.1093/rap/rkab009. eCollection 2021. PMID 33748660
- [Derived] Menter A, Cather JC, Jarratt M, Meng X, Guana A, Nyirady J. Efficacy of Secukinumab on Moderate-to-severe Plaque Psoriasis Affecting Different Body Regions: a Pooled Analysis of Four Phase 3 Studies. Dermatol Ther (Heidelb). 2016 Dec;6(4):639-647. doi: 10.1007/s13555-016-0140-7. Epub 2016 Aug 30. PMID 27576559
- [Derived] Kircik L, Fowler J, Weiss J, Meng X, Guana A, Nyirady J. Efficacy of Secukinumab for Moderate-to-Severe Head and Neck Psoriasis Over 52 Weeks: Pooled Analysis of Four Phase 3 Studies. Dermatol Ther (Heidelb). 2016 Dec;6(4):627-638. doi: 10.1007/s13555-016-0139-0. Epub 2016 Aug 30. PMID 27573260
- [Derived] Gottlieb AB, Langley RG, Philipp S, Sigurgeirsson B, Blauvelt A, Martin R, Papavassilis C, Mpofu S. Secukinumab Improves Physical Function in Subjects With Plaque Psoriasis and Psoriatic Arthritis: Results from Two Randomized, Phase 3 Trials. J Drugs Dermatol. 2015 Aug;14(8):821-33. PMID 26267726
- [Derived] Ohtsuki M, Morita A, Abe M, Takahashi H, Seko N, Karpov A, Shima T, Papavassilis C, Nakagawa H; ERASURE Study Japanese subgroup. Secukinumab efficacy and safety in Japanese patients with moderate-to-severe plaque psoriasis: subanalysis from ERASURE, a randomized, placebo-controlled, phase 3 study. J Dermatol. 2014 Dec;41(12):1039-46. doi: 10.1111/1346-8138.12668. Epub 2014 Oct 30. PMID 25354738
- [Derived] Langley RG, Elewski BE, Lebwohl M, Reich K, Griffiths CE, Papp K, Puig L, Nakagawa H, Spelman L, Sigurgeirsson B, Rivas E, Tsai TF, Wasel N, Tyring S, Salko T, Hampele I, Notter M, Karpov A, Helou S, Papavassilis C; ERASURE Study Group; FIXTURE Study Group. Secukinumab in plaque psoriasis--results of two phase 3 trials. N Engl J Med. 2014 Jul 24;371(4):326-38. doi: 10.1056/NEJMoa1314258. Epub 2014 Jul 9. PMID 25007392
- See also: Plain Language Trial Summaries available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Not all patients that completed Maintenance Period continued in the follow-up Period. Many patients from Maintence rolled into CAIN457A2302E1 study
Period: Induction Period
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo | AIN457 150mg From Placebo | AIN457 300mg From Placebo
Started | 245 | 245 | 248 | 0 | 0
Completed | 230 | 238 | 232 | 0 | 0
Not Completed | 15 | 7 | 16 | 0 | 0
Not completed — Adverse Event | 5 | 3 | 4 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0
Not completed — Protocol deviation | 0 | 1 | 1 | 0 | 0
Not completed — Subject/guardian decision | 9 | 1 | 8 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 0 | 0
Period: Maintenance Period
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo | AIN457 150mg From Placebo | AIN457 300mg From Placebo
Started | 230 | 238 | 18 | 109 | 105
Completed | 201 | 215 | 15 | 100 | 92
Not Completed | 29 | 23 | 3 | 9 | 13
Not completed — Adverse Event | 12 | 5 | 1 | 2 | 4
Not completed — Lack of Efficacy | 10 | 2 | 0 | 2 | 2
Not completed — Lost to Follow-up | 2 | 4 | 0 | 0 | 3
Not completed — Non-compliance with study treatment | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 4 | 0 | 0 | 2
Not completed — Protocol deviation | 1 | 1 | 0 | 0 | 0
Not completed — Subject/guardian decision | 4 | 6 | 2 | 4 | 1
Period: Follow-up Period
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo | AIN457 150mg From Placebo | AIN457 300mg From Placebo
Started | 58 | 47 | 18 | 0 | 0
Completed | 58 | 47 | 18 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo | Total
Number analyzed (Participants) | 245 | 245 | 248 | 738
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (13.33) | 44.9 (13.46) | 45.4 (12.63) | 45.1 (13.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 76 | 76 | 229
  Male | 168 | 169 | 172 | 509

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved >75 or Higher (Psoriasis Area and Severity Index) PASI Score at 12 Weeks
Description: A 75% reduction in the Psoriasis Area and Severity Index (PASI) score (PASI 75) is the current benchmark of primary endpoints for most clinical trials of psoriasis. PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
Time Frame: 12 weeks
Population: Full analysis set (FAS): The FAS was comprised of all patients to whom study treatment had been assigned. Following the intent-to-treat principle, patients were analyzed according to the treatment assigned to at randomization. If the actual stratum was different to the assigned stratum in IRT, the actual stratum was used in analyses.
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 243 | 245 | 246
Percentage of participants | 71.6 | 81.6 | 4.5

2. Primary Outcome: Percentage of Participants Who Achieved (Investigator's Global Assessment) IGA Score of 0 or 1
Description: The IGA mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe. Treatment success was defined as achievement of IGA mod 2001 score of 0 or 1. IGA score of 0 or 1 as an indicator of efficacy.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 244 | 245 | 246
Percentage of Participants | 51.2 | 65.3 | 2.4

3. Secondary Outcome: Percentage of Participants Who Achieved a PASI (Psoriasis Area and Severity Index) Score of 90 or Better at Week 12
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). PASI 90 was defined as participants who achievied ≥ 90% improvement from baseline.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 243 | 245 | 246
Percentage of Participants | 39.1 | 59.2 | 1.2

4. Secondary Outcome: Number of Participants That Maintained the Psoriasis Area and Severity Index (PASI) 75 Response at 52 Weeks of Treatment for Participants Who Were PASI 75 Responders at Week 12
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
Time Frame: 12 and 52 weeks
Population: as for outcome 1
Measure: Number; unit: number of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 245 | 245 | 248
number of participants
  PASI 75 response at Week 12 (n=243, 245, 246) | 174 | 200 | 11
  Maintained PASI 75 response at Wk 52(n=174,200,11) | 126 | 161 | NA — After W12: Efficacy was not focus for PBO group and therefore no data was provided at Week 52

5. Secondary Outcome: Number of Participants That Maintained the IGA Mod 2011 0 or 1 Response at 52 Weeks of Treatment for Participants Who Were IGA Mod 2011 0 or 1 Responders at Week 12
Description: The IGA mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe. Treatment success was defined as achievement of IGA mod 2001 score of 0 or 1.
Time Frame: 12 and 52 weeks
Population: as for outcome 1
Measure: Number; unit: number of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 245 | 245 | 248
number of participants
  IGA mod2011 0or1 response at Wk 12(n=244,245,246) | 125 | 160 | 6
  Maintained IGAmod2011 0or1 resp atWk52 n=125,160,6 | 74 | 119 | NA — After W12: Efficacy was not focus for PBO group and therefore no data was provided at Week 52

6. Secondary Outcome: Change From Baseline to Week 12 in Psoriasis Symptom Diary Items Itching, Pain and Scaling in AIN457 vs Placebo
Description: The Psoriasis Symptom Diary©, a 16-item patient reported outcome (PRO) measure developed and validated in accordance with the FDA PRO Guidance (FDA Guidance for Industry: Patient-Reported Outcome Measures: Use in Medical Product Development to Support Labeling Claims, 2009), demonstrated favorable psychometric properties and usefulness for treatment efficacy evaluation alongside other measures of disease severity in clinical trials for chronic plaque psoriasis.Weekly averages will be derived for each of the 16 questions of the Psoriasis Diary up to Week 12. A weekly average is the sum of the scored item over the course of the study week divided by the number of days on which the item was completed and will be set to missing if four or more daily assessments were missing of the corresponding question. A reduction in score from baseline shows efficacy. Each question has a score of 0 (no symptoms) up to 10 (Severe symptoms)
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 245 | 245 | 248
Scores on a Scale
  itching (n=86,79,84) | -4.86 (0.299) | -545 (0.276) | -0.22 (0.260)
  pain (n=86,79,84) | -3.92 (0.337) | -4.59 (0.322) | 0.06 (0.246)
  scaling (n=86,79,84) | -4.74 (0.307) | -5.49 (0.289) | -0.11 (0.248)

7. Secondary Outcome: Percentage of Participants Achieving PASI 50/75/90/100 Response or IGA 0 or 1 Response up to 12 Weeks Induction Period
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (max). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). PASI 50, 75, 90 and 100 were defined as participants achieving ≥ 50%, 75%, 90% or 100% improvement from baseline. The IGA mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe.
Time Frame: Week 1,2,3,4,8,12,
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 245 | 245 | 247
Percentage of participants
  Week 1 IGA 0/1 (n=244,245,246) | 0.0 | 0.0 | 0.0
  Week 1 PASI 75 (n=243,245,246) | 0.0 | 0.0 | 0.0
  Week 1 PASI 50 (n=243,245,246) | 2.1 | 4.5 | 0.4
  Week 1 PASI 90 (n=243,245,246) | 0.0 | 0.0 | 0.0
  Week 1 PASI 100 (n=243,245,246) | 0.0 | 0.0 | 0.0
  Week 2 IGA 0/1 n=244,245,246) | 1.2 | 4.5 | 0.0
  Week 2 PASI 75 (n=243,245,246) | 0.8 | 4.1 | 0.0
  Week 2 PASI 50 (n=243,245,246) | 18.5 | 28.2 | 3.3
  Week 2 PASI 90 (n=243,245,246) | 0.0 | 0.8 | 0.0
  Week 2 PASI 100 (n=243,245,246) | 0.0 | 0.0 | 0.0
  Week 3 IGA 0/1( n=244,245,246) | 6.6 | 11.0 | 0.4
  Week 3 PASI 75 (n=243,245,246) | 8.2 | 15.5 | 1.2
  Week 3 PASI 50 (n=243,245,246) | 41.2 | 53.1 | 4.9
  Week 3 PASI 90 (n=243,245,246) | 0.8 | 2.9 | 0.0
  Week 3 PASI 100 (n=243,245,246) | 0.0 | 0.8 | 0.0
  Week 4 IGA 0/1( n=244,245,246) | 17.2 | 26.1 | 1.2
  Week 4 PASI 75 (n=243,245,246) | 24.3 | 38.0 | 0.8
  Week 4 PASI 50 (n=243,245,246) | 63.0 | 74.7 | 7.3
  Week 4 PASI 90 (n=243,245,246) | 5.8 | 10.6 | 0.4
  Week 4 PASI 100 (n=243,245,246) | 0.8 | 3.7 | 0.0
  Week 8 IGA 0/1( n=244,245,246) | 42.2 | 60.0 | 1.6
  Week 8 PASI 75 (n=243,245,246) | 61.7 | 76.7 | 2.8
  Week 8 PASI 50 (n=243,245,246) | 88.5 | 92.2 | 9.3
  Week 8 PASI 90 (n=243,245,246) | 28.8 | 47.8 | 1.2
  Week 8 PASI 100 (n=243,245,246) | 8.2 | 16.7 | 0.0
  Week 12 IGA 0/1( n=244,245,246) | 51.2 | 65.3 | 2.4
  Week 12 PASI 75 (n=243,245,246) | 71.6 | 81.6 | 4.5
  Week 12 PASI 50 (n=243,245,246) | 83.5 | 90.6 | 8.9
  Week 12 PASI 90 (n=243,245,246) | 39.1 | 59.2 | 1.2
  Week 12 PASI 100 (n=243,245,246) | 12.8 | 28.6 | 0.8

8. Secondary Outcome: Percentage of Participants Achieving PASI 50/75/90/100 Response or IGA 0 or 1 Response Maintenance Period After Week 12 to Week 52
Description: as for outcome 7
Time Frame: Week 13,14,15,16,20,24,28,32,36,40,44,48,52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo | AIN457 150mg From Placebo | AIN457 300mg From Placebo
Number analyzed (Participants) | 245 | 245 | 18 | 108 | 105
Percentage of participants
  Week 13 IGA 0/1 (n=244,245,18, 108, 104) | 51.6 | 66.9 | 33.3 | 0.9 | 1.9
  Week 13 PASI 75 (n=243,245,18, 108, 104) | 70.8 | 79.6 | 55.6 | 2.8 | 0.0
  Week 13 PASI 50 (n=243,245,18, 108, 104) | 81.5 | 87.3 | 77.8 | 12.0 | 13.5
  Week 13 PASI 90 (n=243,245,18, 108, 104) | 44.9 | 60.8 | 22.2 | 0.9 | 0.0
  Week 13 PASI 100 (n=243,245,18, 108, 104) | 14.0 | 30.2 | 11.1 | 0.0 | 0.0
  Week 14 IGA 0/1 (n=244,245,18, 108, 104) | 55.3 | 74.7 | 33.3 | 4.6 | 10.6
  Week 14 PASI 75 (n=243,245,18, 108, 104) | 72.0 | 86.1 | 55.6 | 7.4 | 14.4
  Week 14 PASI 50 (n=243,245,18, 108, 104) | 83.1 | 91.4 | 83.3 | 34.3 | 38.5
  Week 14 PASI 90 (n=243,245,18, 108, 104) | 48.6 | 68.2 | 27.8 | 0.9 | 0.0
  Week 14 PASI 100 (n=243,245,18, 108, 104) | 16.5 | 35.5 | 11.1 | 0.0 | 0.0
  Week 15 IGA 0/1 (n=244,245,18, 108, 104) | 57.4 | 75.1 | 33.3 | 13.0 | 19.2
  Week 15 PASI 75 (n=243,245,18, 108, 104) | 75.3 | 87.8 | 55.6 | 13.9 | 26.9
  Week 15 PASI 50 (n=243,245,18, 108, 104) | 86.4 | 92.2 | 72.2 | 55.6 | 66.3
  Week 15 PASI 90 (n=243,245,18, 108, 104) | 51.0 | 68.6 | 27.8 | 2.8 | 6.7
  Week 15 PASI 100 (n=243,245,18, 108, 104) | 19.8 | 40.8 | 11.1 | 0.0 | 0.0
  Week 16 IGA 0/1 (n=244,245,18, 108, 104) | 58.2 | 73.5 | 38.9 | 25.9 | 30.8
  Week 16 PASI 75 (n=243,245,18, 108, 104) | 77.4 | 86.1 | 61.1 | 33.3 | 47.1
  Week 16 PASI 50 (n=243,245,18, 108, 104) | 87.2 | 91.4 | 77.8 | 68.5 | 81.7
  Week 16 PASI 90 (n=243,245,18, 108, 104) | 53.5 | 69.8 | 33.3 | 10.2 | 15.4
  Week 16 PASI 100 (n=243,245,18, 108, 104) | 21.0 | 41.6 | 22.2 | 0.9 | 4.8
  Week 20 IGA 0/1 (n=244,245,18, 108, 104) | 57.4 | 74.7 | 38.9 | 51.9 | 55.8
  Week 20 PASI 75 (n=243,245,18, 108, 104) | 77.0 | 86.9 | 72.2 | 66.7 | 75.0
  Week 20 PASI 50 (n=243,245,18, 108, 104) | 89.3 | 92.7 | 88.9 | 87.0 | 91.3
  Week 20 PASI 90 (n=243,245,18, 108, 104) | 51.9 | 69.8 | 38.9 | 38.0 | 50.0
  Week 20 PASI 100 (n=243,245,18, 108, 104) | 21.8 | 43.3 | 16.7 | 5.6 | 19.2
  Week 24 IGA 0/1 (n=244,245,18, 108, 104) | 58.2 | 71.4 | 50.0 | 57.4 | 72.1
  Week 24 PASI 75 (n=243,245,18, 108, 104) | 77.8 | 85.7 | 66.7 | 76.9 | 81.7
  Week 24 PASI 50 (n=243,245,18, 108, 104) | 86.8 | 91.0 | 88.9 | 91.7 | 93.3
  Week 24 PASI 90 (n=243,245,18, 108, 104) | 54.7 | 70.2 | 38.9 | 50.9 | 62.5
  Week 24 PASI 100 (n=243,245,18, 108, 104) | 23.9 | 42.4 | 16.7 | 16.7 | 26.0
  Week 28 IGA 0/1 (n=244,245,18, 108, 104) | 53.7 | 68.6 | 50.0 | 61.1 | 76.0
  Week 28 PASI 75 (n=243,245,18, 108, 104) | 72.4 | 82.9 | 72.2 | 74.1 | 87.5
  Week 28 PASI 50 (n=243,245,18, 108, 104) | 84.4 | 90.2 | 83.3 | 91.7 | 93.3
  Week 28 PASI 90 (n=243,245,18, 108, 104) | 53.1 | 68.6 | 50.0 | 50.0 | 71.2
  Week 28 PASI 100 (n=243,245,18, 108, 104) | 24.3 | 43.3 | 16.7 | 24.1 | 33.7
  Week 32 IGA 0/1 (n=244,245,18, 108, 104) | 50.8 | 68.2 | 44.4 | 57.4 | 76.0
  Week 32 PASI 75 (n=243,245,18, 108, 104) | 72.0 | 81.2 | 61.1 | 75.0 | 89.4
  Week 32 PASI 50 (n=243,245,18, 108, 104) | 86.4 | 88.6 | 77.8 | 88.9 | 94.2
  Week 32 PASI 90 (n=243,245,18, 108, 104) | 48.1 | 68.2 | 44.4 | 50.9 | 70.2
  Week 32 PASI 100 (n=243,245,18, 108, 104) | 22.2 | 43.7 | 16.7 | 22.2 | 39.4
  Week 36 IGA 0/1 (n=244,245,18, 108, 104) | 48.0 | 66.9 | 38.9 | 60.2 | 70.2
  Week 36 PASI 75 (n=243,245,18, 108, 104) | 67.5 | 79.2 | 61.1 | 73.1 | 86.5
  Week 36 PASI 50 (n=243,245,18, 108, 104) | 80.2 | 86.9 | 88.9 | 88.9 | 89.4
  Week 36 PASI 90 (n=243,245,18, 108, 104) | 44.4 | 67.3 | 44.4 | 52.8 | 64.4
  Week 36 PASI 100 (n=243,245,18, 108, 104) | 22.2 | 42.4 | 16.7 | 25.0 | 43.3
  Week 40 IGA 0/1 (n=244,245,18, 108, 104) | 47.1 | 64.9 | 44.4 | 57.4 | 69.2
  Week 40 PASI 75 (n=243,245,18, 108, 104) | 65.4 | 76.7 | 66.7 | 69.4 | 81.7
  Week 40 PASI 50 (n=243,245,18, 108, 104) | 78.6 | 84.9 | 83.3 | 88.0 | 88.5
  Week 40 PASI 90 (n=243,245,18, 108, 104) | 44.0 | 64.9 | 44.4 | 50.9 | 65.4
  Week 40 PASI 100 (n=243,245,18, 108, 104) | 21.0 | 40.8 | 27.8 | 24.1 | 42.3
  Week 44 IGA 0/1 (n=244,245,18, 108, 104) | 44.3 | 60.4 | 44.4 | 57.4 | 72.1
  Week 44 PASI 75 (n=243,245,18, 108, 104) | 63.4 | 79.2 | 61.1 | 68.5 | 79.8
  Week 44 PASI 50 (n=243,245,18, 108, 104) | 77.4 | 84.5 | 83.3 | 89.8 | 89.4
  Week 44 PASI 90 (n=243,245,18, 108, 104) | 42.8 | 61.2 | 38.9 | 47.2 | 66.3
  Week 44 PASI 100 (n=243,245,18, 108, 104) | 21.8 | 37.1 | 11.1 | 23.1 | 38.5
  Week 48 IGA 0/1 (n=244,245,18, 108, 104) | 41.4 | 62.9 | 27.8 | 50.0 | 69.2
  Week 48 PASI 75 (n=243,245,18, 108, 104) | 62.1 | 77.6 | 66.7 | 68.5 | 76.9
  Week 48 PASI 50 (n=243,245,18, 108, 104) | 77.4 | 84.9 | 83.3 | 86.1 | 83.7
  Week 48 PASI 90 (n=243,245,18, 108, 104) | 39.5 | 63.7 | 38.9 | 45.4 | 63.5
  Week 48 PASI 100 (n=243,245,18, 108, 104) | 22.2 | 40.4 | 11.1 | 20.4 | 37.5
  Week 52 IGA 0/1 (n=244,245,18, 108, 104) | 73.4 | 87.3 | 38.9 | 76.9 | 66.3
  Week 52 PASI 75 (n=243,245,18, 108, 104) | 86.8 | 94.3 | 66.7 | 88.0 | 73.1
  Week 52 PASI 50(n=243,245,18, 108, 104) | 91.8 | 95.9 | 83.3 | 96.3 | 81.7
  Week 52 PASI 90 (n=243,245,18, 108, 104) | 73.3 | 84.5 | 33.3 | 66.7 | 62.5
  Week 52 PASI 100 (n=243,245,18, 108, 104) | 41.2 | 62.0 | 11.1 | 36.1 | 43.3

9. Secondary Outcome: Mean Percent Change From Baseline in PASI Scores up to Week 12 - Induction Period
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). A negative mean percentage change indicates improvement.
Time Frame: Baseline, Week 1,2,3,4,8,12,
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 245 | 245 | 247
Percent Change
  Week 1 (n=243,243,242) | -12.08 (19.225) | -17.50 (17.317) | -3.70 (14.756)
  Week 2 (n=243,245,243) | -28.61 (21.982) | -36.51 (21.850) | -5.63 (23.616)
  Week 3 (n=243,245,243) | -42.79 (23.695) | -51.59 (22.415) | -8.62 (25.785)
  Week 4 (n=243,245,245) | -55.73 (24.252) | -64.61 (22.080) | -8.89 (28.165)
  Week 8 (n=243,245,245) | -76.35 (20.427) | -82.98 (19.331) | -8.15 (32.755)
  Week 12 (n=243,245,245) | -80.87 (20.512) | -87.72 (17.729) | -5.89 (36.606)

10. Secondary Outcome: Mean Percent Change From Baseline in PASI Scores Maintenance Period After Week 12 to Week 52
Description: as for outcome 9
Time Frame: Week 13,14,15,16,20,24,28,32,36,40,44,48,52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo | AIN457 150mg From Placebo | AIN457 300mg From Placebo
Number analyzed (Participants) | 245 | 245 | 18 | 108 | 105
Percent change
  Week 13 (n=243,245,18,102,96) | -83.12 (19.313) | -89.55 (15.935) | -63.10 (36.827) | -21.03 (28.240) | -21.66 (29.891)
  Week 14 (n=243,245,18,107,102) | -84.47 (18.832) | -90.83 (15.013) | -68.74 (30.225) | -39.20 (26.228) | -41.97 (28.809)
  Week 15 (n=243,245,18,107,103) | -84.67 (19.407) | -91.40 (14.769) | -67.15 (32.972) | -51.78 (23.561) | -57.77 (23.166)
  Week 16 (n=243,245,18,107,103) | -85.20 (19.213) | -91.37 (15.367) | -73.38 (28.051) | -62.19 (23.591) | -70.15 (20.686)
  Week 20 (n=243,245,18,107,103) | -85.75 (17.904) | -90.86 (16.263) | -80.57 (22.454) | -77.75 (20.587) | -84.53 (16.030)
  Week 24 (n=243,245,18,107,103) | -85.46 (20.240) | -90.83 (16.652) | -78.06 (25.062) | -83.19 (18.635) | -89.20 (13.969)
  Week 28 (n=243,245,18,107,103) | -84.72 (20.417) | -90.15 (17.600) | -79.55 (23.943) | -84.07 (19.819) | -91.24 (11.849)
  Week 32 (n=243,245,18,107,103) | -83.98 (21.887) | -89.90 (17.775) | -75.94 (25.879) | -84.26 (20.622) | -91.09 (13.240)
  Week 36(n=243,245,18,107,103) | -81.87 (25.048) | -90.04 (17.981) | -78.37 (24.608) | -83.68 (20.328) | -89.97 (16.373)
  Week 40(n=243,245,18,107,103) | -81.37 (25.395) | -89.62 (17.385) | -78.32 (24.770) | -82.83 (20.762) | -89.76 (17.029)
  Week 44 (n=243,245,18,107,103) | -80.81 (25.651) | -88.97 (17.804) | -79.96 (22.354) | -83.44 (18.277) | -89.37 (17.176)
  Week 48(n=243,245,18,107,103) | -79.78 (26.471) | -89.35 (17.281) | -79.54 (21.506) | -83.40 (18.736) | -88.44 (18.083)
  Week 52 (n=243,245,18,107,103) | -79.74 (26.524) | -88.42 (19.132) | -79.64 (22.169) | -82.14 (18.554) | -87.66 (20.615)

11. Secondary Outcome: Percentage of Participants in Each IGA Mod 2011 Score Category up to Week 12 - Induction Period
Description: The IGA mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe.
Time Frame: Baseline, Week 1,2,3,4,8,12,
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 245 | 245 | 247
Percentage of participants
  Week 1 (n=244,243,243) clear | 0.0 (19.225) | 0.0 (17.317) | 0.0 (14.756)
  Week 1 (n=244,243,243) almost clear | 0.0 (21.982) | 0.0 (21.850) | 0.0 (23.616)
  Week 1 (n=244,243,243) mild | 6.6 (23.695) | 9.1 (22.415) | 4.1 (25.785)
  Week 1 (n=244,243,243) moderate | 66.4 (24.252) | 68.7 (22.080) | 60.9 (28.165)
  Week 1 (n=244,243,243) severe | 27.0 | 22.2 | 35.0
  Week 2 (n=244,245,244) clear | 0.0 | 0.0 | 0.0
  Week 2 (n=244,245,244) almost clear | 1.2 | 4.5 | 0.0
  Week 2 (n=244,245,244) mild | 23.0 | 27.8 | 5.3
  Week 2 (n=244,245,244) moderate | 57.0 | 55.5 | 59.8
  Week 2 (n=244,245,244) severe | 18.9 | 12.2 | 34.8
  Week 3 (n=244,245,244) clear | 0.0 | 1.2 | 0.0
  Week 3 (n=244,245,244) almost clear | 6.6 | 9.8 | 0.4
  Week 3 (n=244,245,244) mild | 34.0 | 43.3 | 7.0
  Week 3 (n=244,245,244) moderate | 49.2 | 40.4 | 58.6
  Week 3 (n=244,245,244) severe | 10.2 | 5.3 | 34.0
  Week 4 (n=244,245,246) clear | 0.4 | 3.7 | 0.0
  Week 4 (n=244,245,246) almost clear | 16.8 | 22.9 | 1.6
  Week 4 (n=244,245,246) mild | 40.2 | 43.7 | 7.3
  Week 4 (n=244,245,246) moderate | 37.3 | 26.5 | 58.1
  Week 4 (n=244,245,246) severe | 5.3 | 3.3 | 32.9
  Week 8 (n=244,245,246) clear | 10.2 | 20.4 | 0.0
  Week 8 (n=244,245,246) almost clear | 32.0 | 39.6 | 1.6
  Week 8 (n=244,245,246) mild | 38.9 | 29.0 | 8.1
  Week 8 (n=244,245,246) moderate | 16.4 | 10.2 | 53.3
  Week 8 (n=244,245,246) severe | 2.5 | 0.8 | 37.0
  Week 12 (n=244,245,246) clear | 16.4 | 32.2 | 0.8
  Week 12 (n=244,245,246) almost clear | 38.5 | 36.3 | 1.6
  Week 12 (n=244,245,246) mild | 29.1 | 23.3 | 6.5
  Week 12 (n=244,245,246) moderate | 14.8 | 6.9 | 55.3
  Week 12 (n=244,245,246) severe | 1.2 | 1.2 | 35.8

12. Secondary Outcome: Percentage of Participants in Each IGA Mod 2011 Score Category Maintenance Period After Week 12 to Week 52
Description: as for outcome 11
Time Frame: Week 13,14,15,16,20,24,28,32,36,40,44,48,52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo | AIN457 150mg From Placebo | AIN457 300mg From Placebo
Number analyzed (Participants) | 245 | 245 | 18 | 108 | 105
Percentage of participants
  Week 13 (n=244,245,18,103,96) clear | 17.6 (19.313) | 38.0 (15.935) | 11.1 (36.827) | 0.0 (28.240) | 0.0 (29.891)
  Week 13 (n=244,245,18,103,96) almost clear | 40.6 (18.832) | 35.9 (15.013) | 22.2 (30.225) | 1.0 (26.228) | 2.1 (28.809)
  Week 13 (n=244,245,18,103,96) mild | 27.0 (19.407) | 19.2 (14.769) | 27.8 (32.972) | 15.5 (23.561) | 14.6 (23.166)
  Week 13 (n=244,245,18,103,96) moderate | 12.7 (19.213) | 6.5 (15.367) | 27.8 (28.051) | 61.2 (23.591) | 59.4 (20.686)
  Week 13 (n=244,245,18,103,96) severe | 2.0 (17.904) | 0.4 (16.263) | 11.1 (22.454) | 22.3 (20.587) | 24.0 (16.030)
  Week 14 (n=244,245,18,108,102) clear | 19.3 (20.240) | 41.6 (16.652) | 16.7 (25.062) | 0.0 (18.635) | 0.0 (13.969)
  Week 14 (n=244,245,18,108,102)almost clear | 42.3 (20.417) | 36.7 (17.600) | 16.7 (23.943) | 4.6 (19.819) | 10.8 (11.849)
  Week 14 (n=244,245,18,108,102) mild | 25.0 (21.887) | 13.5 (17.775) | 33.3 (25.879) | 30.6 (20.622) | 27.5 (13.240)
  Week 14 (n=244,245,18,108,102)moderate | 12.3 (25.048) | 7.3 (17.981) | 22.2 (24.608) | 56.5 (20.328) | 50.0 (16.373)
  Week 14 (n=244,245,18,108,102)severe | 1.2 (25.395) | 0.8 (17.385) | 11.1 (24.770) | 8.3 (20.762) | 11.8 (17.029)
  Week 15 (n=244,245,18,108,103) clear | 22.1 (25.651) | 45.3 (17.804) | 11.1 (22.354) | 0.0 (18.277) | 1.9 (17.176)
  Week 15 (n=244,245,18,108,103) almost clear | 38.9 (26.471) | 33.9 (17.281) | 22.2 (21.506) | 13.9 (18.736) | 17.5 (18.083)
  Week 15 (n=244,245,18,108,103) mild | 27.5 (26.524) | 14.7 (19.132) | 33.3 (22.169) | 38.9 (18.554) | 39.8 (20.615)
  Week 15 (n=244,245,18,108,103) moderate | 10.2 | 5.3 | 22.2 | 42.6 | 35.9
  Week 15 (n=244,245,18,108,103) severe | 1.2 | 0.8 | 11.1 | 4.6 | 4.9
  Week 16 (n=244,245,18,108,103) clear | 23.8 | 47.3 | 22.2 | 0.0 | 6.8
  Week 16 (n=244,245,18,108,103) almost clear | 37.7 | 30.6 | 16.7 | 0.0 | 24.3
  Week 16 (n=244,245,18,108,103) mild | 26.6 | 15.9 | 27.8 | 7.4 | 39.8
  Week 16 (n=244,245,18,108,103) moderate | 10.7 | 5.3 | 22.2 | 57.4 | 26.2
  Week 16 (n=244,245,18,108,103) severe | 1.2 | 0.8 | 11.1 | 35.2 | 2.9
  Week 20 (n=244,245,18,108,103) clear | 23.8 | 46.1 | 16.7 | 0.0 | 26.2
  Week 20 (n=244,245,18,108,103) almost clear | 37.3 | 31.8 | 22.2 | 1.0 | 31.1
  Week 20 (n=244,245,18,108,103) mild | 26.2 | 14.3 | 33.3 | 15.5 | 32.0
  Week 20 (n=244,245,18,108,103) moderate | 11.5 | 7.3 | 16.7 | 61.2 | 10.7
  Week 20 (n=244,245,18,108,103) severe | 1.2 | 0.4 | 11.1 | 22.3 | 0.0
  Week 24 (n=244,245,18,108,103) clear | 27.0 | 46.5 | 16.7 | 0.0 | 32.0
  Week 24 (n=244,245,18,108,103) almost clear | 35.7 | 29.0 | 33.3 | 4.6 | 41.7
  Week 24 (n=244,245,18,108,103) mild | 24.6 | 15.1 | 22.2 | 30.6 | 20.4
  Week 24 (n=244,245,18,108,103) moderate | 10.7 | 7.8 | 16.7 | 56.5 | 5.8
  Week 24 (n=244,245,18,108,103) severe | 2.0 | 1.6 | 11.1 | 8.3 | 0.0
  Week 28 (n=244,245,18,108,103) clear | 26.6 | 46.5 | 11.1 | 0.0 | 38.8
  Week 28 (n=244,245,18,108,103) almost clear | 32.8 | 26.5 | 38.9 | 13.9 | 40.8
  Week 28 (n=244,245,18,108,103) mild | 25.8 | 16.7 | 16.7 | 38.9 | 14.6
  Week 28 (n=244,245,18,108,103) moderate | 12.7 | 9.4 | 27.8 | 42.6 | 5.8
  Week 28 (n=244,245,18,108,103) severe | 2.0 | 0.8 | 5.6 | 4.6 | 0.0
  Week 32 (n=244,245,18,108,103) clear | 26.2 | 46.5 | 16.7 | 29.6 | 42.7
  Week 32 (n=244,245,18,108,103) almost clear | 30.3 | 26.5 | 27.8 | 30.6 | 35.9
  Week 32 (n=244,245,18,108,103) mild | 27.0 | 16.7 | 27.8 | 22.2 | 13.6
  Week 32 (n=244,245,18,108,103) moderate | 14.3 | 9.0 | 22.2 | 14.8 | 7.8
  Week 32 (n=244,245,18,108,103) severe | 2.0 | 1.2 | 5.6 | 2.8 | 0.0
  Week 36 (n=244,245,18,108,103) clear | 28.3 | 46.5 | 11.1 | 28.7 | 45.6
  Week 36 (n=244,245,18,108,103) almost clear | 27.0 | 26.9 | 27.8 | 33.3 | 29.1
  Week 36 (n=244,245,18,108,103) mild | 25.4 | 16.7 | 33.3 | 18.5 | 16.5
  Week 36 (n=244,245,18,108,103) moderate | 16.8 | 8.2 | 16.7 | 16.7 | 8.7
  Week 36 (n=244,245,18,108,103) severe | 2.5 | 1.6 | 11.1 | 2.8 | 0.0
  Week 40 (n=244,245,18,108,103) clear | 28.7 | 46.1 | 22.2 | 25.9 | 44.7
  Week 40 (n=244,245,18,108,103) almost clear | 25.8 | 25.3 | 22.2 | 34.3 | 31.1
  Week 40 (n=244,245,18,108,103) mild | 25.0 | 17.1 | 27.8 | 21.3 | 11.7
  Week 40 (n=244,245,18,108,103) moderate | 18.4 | 10.2 | 16.7 | 15.7 | 11.7
  Week 40 (n=244,245,18,108,103) severe | 2.0 | 1.2 | 11.1 | 2.8 | 1.0
  Week 44 (n=244,245,18,108,103) clear | 27.5 | 42.9 | 5.6 | 25.9 | 40.8
  Week 44 (n=244,245,18,108,103) almost clear | 25.0 | 24.1 | 38.9 | 33.3 | 36.9
  Week 44 (n=244,245,18,108,103) mild | 25.4 | 20.4 | 22.2 | 20.4 | 8.7
  Week 44 (n=244,245,18,108,103) moderate | 20.1 | 11.8 | 27.8 | 17.6 | 11.7
  Week 44 (n=244,245,18,108,103) severe | 2.0 | 0.8 | 5.6 | 2.8 | 1.9
  Week 48 (n=244,245,18,108,103) clear | 27.0 | 44.5 | 11.1 | 25.9 | 43.7
  Week 48 (n=244,245,18,108,103) almost clear | 22.1 | 25.3 | 16.7 | 28.7 | 34.0
  Week 48 (n=244,245,18,108,103) mild | 27.9 | 16.3 | 50.0 | 27.8 | 9.7
  Week 48 (n=244,245,18,108,103) moderate | 20.1 | 12.7 | 16.7 | 14.8 | 11.7
  Week 48 (n=244,245,18,108,103) severe | 2.9 | 1.2 | 5.6 | 2.8 | 1.0
  Week 52 (n=244,245,18,108,103) clear | 25.8 | 43.3 | 11.1 | 21.3 | 44.7
  Week 52 (n=244,245,18,108,103) almost clear | 24.2 | 24.1 | 27.8 | 31.5 | 29.1
  Week 52 (n=244,245,18,108,103) mild | 29.1 | 19.6 | 27.8 | 28.7 | 12.6
  Week 52 (n=244,245,18,108,103) moderate | 16.0 | 11.4 | 27.8 | 15.7 | 11.7
  Week 52 (n=244,245,18,108,103) severe | 4.9 | 1.6 | 5.6 | 2.8 | 1.9

13. Secondary Outcome: Time to PASI 75 Response up to 12 Weeks
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (max). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). PASI 75 was defined as participants achieving ≥ 75% improvement from baseline.
Time Frame: Week 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 245 | 245 | 247
days | 57 [55 to 85] | 57 [29 to 59] | NA [NA to NA] — median could not be calculated because less than 50% of the participants achieved PASI 75

14. Secondary Outcome: Mean Percent Change From Baseline in EuroQOL 5-Dimension Health Status Questionnaire (EQ-5D) Health State Assessment (From 0 to 100) Induction Period
Description: The EQ-5D is an instrument used to assess a participant's health status. The instrument includes a descriptive profile and a visual analog scale (VAS). The descriptive profile includes 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension had 3 response levels: no problems, some problems and severe problems. The VAS is a vertical scale that assesses the health status from 0 (worst possible health state) to 100 (best possible health state). This outcome measures the percent change in VAS score. Positive mean percent changes indicate improvement.
Time Frame: Baseline, Week 4,8, 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 245 | 245 | 247
percent change
  Week 4 (238, 236,235) | 38.1 (95.93) [55 to 85] | 57.1 (234.10) [29 to 59] | 6.3 (59.30) [NA to NA]
  Week 8 (241, 242,241) | 52.3 (142.28) | 72.7 (306.36) | 6.3 (65.47)
  Week 12 (242, 242,242) | 58.5 (158.66) | 76.3 (281.48) | 5.4 (67.60)

15. Secondary Outcome: Mean Percent Change From Baseline in EuroQOL 5-Dimension Health Status Questionnaire (EQ-5D) Health State Assessment (From 0 to 100) Maintenance Period
Description: as for outcome 14
Time Frame: Week 12, 24, 36, 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo | AIN457 150mg From Placebo | AIN457 300mg From Placebo
Number analyzed (Participants) | 245 | 245 | 18 | 108 | 105
Percent Change
  Week 12 (242, 242,18, 108, 104) | 58.5 (158.66) | 76.3 (281.48) | 37.7 (83.41) | -0.1 (38.95) | 3.3 (79.45)
  Week 24 (242, 242,18, 108, 97) | 55.8 (140.46) | 78.0 (299.91) | 48.1 (92.06) | 28.1 (55.71) | 39.7 (80.03)
  Week 36 (242, 242,18, 108, 100) | 55.1 (129.87) | 80.5 (300.89) | 45.3 (77.11) | 28.5 (60.39) | 43.8 (100.57)
  Week 52 (242, 242,18, 108,100) | 54.3 (128.86) | 76.9 (299.07) | 43.9 (81.50) | 28.3 (60.68) | 41.3 (95.90)

16. Secondary Outcome: Percentage Changes in the Dermatology Life Quality Index (DLQI) During Induction Period
Description: The DLQI is a ten item general dermatology disability index designed to assess health-related quality of life in adult participants with skin diseases such as eczema, psoriasis, acne and viral worts. It is a self-administered questionnaire which includes domains of daily activity, leisure, personal relationships, symptoms and feelings, treatment and school/work activities. Each domain has 4 response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is a valid score also and is scored as 0. The DLQI total score is a sum of all 10 responses. Scores range from 0 to 30 with higher scores indicating greater health-related quality of life impairment. A negative mean percentage change from baseline indicates improvement.
Time Frame: Baseline, Week 4, 8 & 12
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Percent Change
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 245 | 245 | 247
Percent Change
  Week 4 (n=237,236,232) | -55.0 [-58.9 to -50.7] | -62.5 [-66.7 to -58.6] | -5.0 [-10.1 to 0.0]
  Week 8 (n=241,242,239) | -73.1 [-76.7 to -69.2] | -81.5 [-84.4 to -79.0] | -8.3 [-13.3 to -2.6]
  Week 12 (n=242,242,240) | -77.8 [-81.3 to -75.0] | -86.4 [-88.9 to -83.3] | -9.1 [-15.6 to -3.3]

17. Secondary Outcome: Percentage Changes in the Dermatology Life Quality Index (DLQI) During Maintenance Period
Description: as for outcome 16
Time Frame: Week 12,24, 36 & 52
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Percent Change
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo | AIN457 150mg From Placebo | AIN457 300mg From Placebo
Number analyzed (Participants) | 245 | 245 | 18 | 108 | 105
Percent Change
  Week 12 (242,242,17,108,104) | -77.8 [-81.3 to -75.0] | -86.4 [-88.9 to -83.3] | -58.3 [-80.0 to -41.7] | -7.1 [-16.7 to 3.4] | -4.4 [-13.9 to 3.4]
  Week 24 (242,242,17,108,97) | -83.3 [-87.5 to -79.4] | -89.6 [-92.5 to -86.0] | -76.6 [-88.9 to -59.6] | -83.3 [-87.5 to -76.7] | -83.3 [-89.9 to -76.6]
  Week 36 (242,242,17,108,100) | -78.6 [-83.3 to -75.0] | -91.7 [-94.2 to -88.9] | -77.9 [-93.3 to -47.2] | -78.5 [-85.7 to -66.7] | -90.0 [-93.3 to -82.7]
  Week 52 (242,242,17,108,100) | -76.5 [-80.6 to -72.3] | -88.9 [-92.3 to -85.7] | -64.4 [-83.3 to -12.5] | -75.0 [-82.8 to -66.2] | -88.9 [-92.9 to -82.9]

18. Secondary Outcome: Percentage of Participants Who Achieved Dermatology Life Quality Index (DLQI) of 0 or 1 During Induction Period
Description: as for outcome 16
Time Frame: Week 4, 8, 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 245 | 245 | 247
Percentage of Participants
  Week 4 (238, 237, 235) | 17.6 | 23.6 | 6.4
  Week 8 (242,243,241) | 39.7 | 48.1 | 10.0
  Week 12 (243,243,243) | 46.1 | 58.8 | 10.3

19. Secondary Outcome: Percentage of Participants Who Achieved Dermatology Life Quality Index (DLQI) of 0 or 1 During Maintenance Period
Description: as for outcome 16
Time Frame: Week 12,24,36, & 52
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo | AIN457 150mg From Placebo | AIN457 300mg From Placebo
Number analyzed (Participants) | 245 | 245 | 18 | 108 | 105
Percentage of Participants
  Week 12 (243,243,18,108,105) | 46.1 | 58.8 | 27.8 | 10.2 | 8.6
  Week 24 (243,243,18,108,98) | 54.7 | 64.6 | 50.0 | 53.7 | 67.3
  Week 36 (243,243,18,108,101) | 51.9 | 68.7 | 50.0 | 56.5 | 69.3
  Week 52 (243,243,18,108,101) | 48.6 | 66.3 | 22.2 | 52.8 | 67.3

20. Secondary Outcome: Percentage of Participants Achieving PASI 75, PASI 90 and IGA Mod 2011 0 or 1 Response at Week 12 by Previous Exposure to Biologic Systemic Therapy or Anti-TNF-α Therapy and Failed to Respond to a Previous Biologic or Anti-TNF-α Therapy Psoriasis Therapy
Description: PASI is an assessment of lesion severity & affected area into a single score:0(no disease)to 72(max. disease).Body is divided into 4 areas for scoring(head,arms,trunk,legs)each area is scored separately & then added for final PASI.For each area, % of skin involved is estimated:0(0%)to 6(90-100%)& severity is estimated by clinical signs, erythema,induration & desquamation;scale 0(none) to 4(max). Final PASI=sum of severity parameters for each area* area score weight of section(head:0.1,arms:0.2 body:0.3 legs:0.4).PASI 75, 90 is patients achieving≥75%or90% improvement from baseline.The IGA mod 2011 scale is static, exclusively to the patients disease at assessment,& not with any of the patient's previous disease states at other visits.The scores are:0=clear,1=almost clear,2= mild,3=moderate&4=severe.Response variables PASI 75,90, IGA mod 2011 0 or 1 response at wk 12 was scored versus previous psoriasis systemic therapy & response to previous biologic systemic therapy by treatment
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 245 | 245 | 247
Percentage of participants
  IGA 0/1 biologic (29, 19, 24) | 41.4 | 57.9 | 4.2
  PASI 75 biologic (29, 19, 24) | 48.3 | 57.9 | 12.5
  PASI 90 biologic (29, 19, 24) | 24.1 | 31.6 | 4.2
  IGA 0/1 anti-TNF-α therapy (18,17,21) | 50.0 | 64.7 | 4.8
  PASI 75 anti-TNF-α therapy (18,17,21) | 55.6 | 64.7 | 14.3
  PASI 90 anti-TNF-α therapy (18,17,21) | 33.3 | 35.3 | 4.8

21. Secondary Outcome: Number of Participants Who Developed Anti-secukinumab Antibodies
Description: The development of anti-secunimubab anti-bodies would decrease a participant's ability to respond to secukinumab treatment.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 245 | 245 | 247
participants | 2 | 0 | 0

ADVERSE EVENTS:
Groups:
- INDUCTION-AIN457 150mg: INDUCTION-AIN457 150mg
- INDUCTION-AIN457 300mg: INDUCTION-AIN457 300mg
- INDUCTION-Placebo: INDUCTION-Placebo
- ENTIRE-AIN457 150mg: ENTIRE-AIN457 150mg
- ENTIRE-AIN457 300mg: ENTIRE-AIN457 300mg
- ENTIRE-Any AIN457 150mg: ENTIRE-Any AIN457 150mg
- ENTIRE-Any AIN457 300mg: ENTIRE-Any AIN457 300mg
- ENTIRE-Placebo: ENTIRE-Placebo
- FOLLOW UP-Any AIN457 150mg: FOLLOW UP-Any AIN457 150mg
- FOLLOW UP-Any AIN457 300mg: FOLLOW UP-Any AIN457 300mg
- FOLLOW UP-Placebo: FOLLOW UP-Placebo
Arm/Group | INDUCTION-AIN457 150mg | INDUCTION-AIN457 300mg | INDUCTION-Placebo | ENTIRE-AIN457 150mg | ENTIRE-AIN457 300mg | ENTIRE-Any AIN457 150mg | ENTIRE-Any AIN457 300mg | ENTIRE-Placebo | FOLLOW UP-Any AIN457 150mg | FOLLOW UP-Any AIN457 300mg | FOLLOW UP-Placebo
Serious Adverse Events (participants affected / at risk) | 4/245 | 6/245 | 4/247 | 15/245 | 17/245 | 19/353 | 19/349 | 5/247 | 1/58 | 1/47 | 0/18
Other Adverse Events (participants affected / at risk) | 108/245 | 102/245 | 77/247 | 172/245 | 161/245 | 228/353 | 229/349 | 85/247 | 8/58 | 8/47 | 5/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INDUCTION-AIN457 150mg (N=245) | INDUCTION-AIN457 300mg (N=245) | INDUCTION-Placebo (N=247) | ENTIRE-AIN457 150mg (N=245) | ENTIRE-AIN457 300mg (N=245) | ENTIRE-Any AIN457 150mg (N=353) | ENTIRE-Any AIN457 300mg (N=349) | ENTIRE-Placebo (N=247) | FOLLOW UP-Any AIN457 150mg (N=58) | FOLLOW UP-Any AIN457 300mg (N=47) | FOLLOW UP-Placebo (N=18)
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ANGINA UNSTABLE (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ABDOMINAL HERNIA OBSTRUCTIVE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PANCREATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
ASTHENIA (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HERNIA (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
BACTERAEMIA (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
PYELONEPHRITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
UROSEPSIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
COMMINUTED FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
CONCUSSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
LARYNGEAL INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
PULMONARY CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
WOUND (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HYPOPROTEINAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
BENIGN NEOPLASM OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
FOLLICULAR THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
CAROTID ARTERY DISSECTION (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HALLUCINATION, AUDITORY (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
PANIC ATTACK (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
OBSTRUCTIVE UROPATHY (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ABORTION INDUCED (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
AORTIC ANEURYSM (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
AORTIC THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | INDUCTION-AIN457 150mg (N=245) | INDUCTION-AIN457 300mg (N=245) | INDUCTION-Placebo (N=247) | ENTIRE-AIN457 150mg (N=245) | ENTIRE-AIN457 300mg (N=245) | ENTIRE-Any AIN457 150mg (N=353) | ENTIRE-Any AIN457 300mg (N=349) | ENTIRE-Placebo (N=247) | FOLLOW UP-Any AIN457 150mg (N=58) | FOLLOW UP-Any AIN457 300mg (N=47) | FOLLOW UP-Placebo (N=18)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 2 | 3 | 0 | 6 | 3 | 6 | 3 | 0 | 0 | 0 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 1 | 1 | 4 | 5 | 4 | 5 | 1 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 4 | 5 | 3 | 9 | 11 | 10 | 16 | 4 | 0 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 1 | 1 | 0 | 6 | 2 | 6 | 4 | 0 | 0 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 5 | 3 | 5 | 1 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 6 | 1 | 6 | 7 | 2 | 8 | 3 | 8 | 0 | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 3 | 2 | 2 | 8 | 4 | 8 | 5 | 2 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 2 | 5 | 2 | 3 | 6 | 4 | 7 | 4 | 0 | 0 | 0
FATIGUE (General disorders) | 8 | 2 | 2 | 9 | 3 | 10 | 3 | 2 | 0 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 3 | 5 | 3 | 15 | 11 | 17 | 14 | 3 | 0 | 0 | 0
ABSCESS LIMB (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 2 | 3 | 1 | 7 | 11 | 8 | 17 | 2 | 0 | 0 | 0
FOLLICULITIS (Infections and infestations) | 4 | 2 | 2 | 10 | 6 | 12 | 9 | 2 | 0 | 0 | 0
FURUNCLE (Infections and infestations) | 1 | 2 | 0 | 5 | 4 | 5 | 4 | 1 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 2 | 1 | 6 | 4 | 7 | 7 | 1 | 0 | 0 | 1
INFLUENZA (Infections and infestations) | 4 | 1 | 2 | 8 | 7 | 8 | 10 | 3 | 1 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 23 | 22 | 19 | 53 | 45 | 69 | 57 | 20 | 1 | 0 | 0
ORAL HERPES (Infections and infestations) | 0 | 3 | 2 | 4 | 6 | 6 | 8 | 2 | 0 | 0 | 0
OTITIS MEDIA (Infections and infestations) | 0 | 3 | 1 | 1 | 6 | 2 | 6 | 1 | 0 | 0 | 0
PERIODONTITIS (Infections and infestations) | 2 | 1 | 1 | 3 | 5 | 3 | 7 | 1 | 0 | 0 | 1
PHARYNGITIS (Infections and infestations) | 2 | 3 | 0 | 8 | 7 | 9 | 9 | 0 | 0 | 0 | 0
RHINITIS (Infections and infestations) | 2 | 2 | 1 | 3 | 6 | 4 | 7 | 1 | 0 | 0 | 0
TINEA PEDIS (Infections and infestations) | 2 | 2 | 0 | 4 | 6 | 8 | 10 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 | 9 | 0 | 28 | 26 | 36 | 32 | 2 | 1 | 0 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 4 | 2 | 6 | 8 | 7 | 11 | 2 | 0 | 0 | 0
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
CONTUSION (Injury, poisoning and procedural complications) | 2 | 5 | 1 | 5 | 5 | 5 | 7 | 1 | 0 | 0 | 0
EXCORIATION (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 2 | 5 | 3 | 7 | 0 | 0 | 0 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2 | 7 | 3 | 8 | 1 | 0 | 0 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 3 | 4 | 0 | 7 | 6 | 8 | 7 | 1 | 0 | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 1 | 5 | 2 | 5 | 0 | 0 | 0 | 0
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 1 | 3 | 2 | 8 | 6 | 13 | 9 | 2 | 0 | 0 | 0
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 5 | 4 | 7 | 0 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 | 2 | 7 | 9 | 9 | 13 | 14 | 8 | 0 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 2 | 4 | 7 | 7 | 9 | 9 | 4 | 0 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 4 | 5 | 5 | 5 | 4 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2 | 6 | 7 | 8 | 8 | 3 | 1 | 0 | 0
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 4 | 6 | 5 | 7 | 4 | 2 | 0 | 0
HEADACHE (Nervous system disorders) | 13 | 12 | 7 | 19 | 22 | 24 | 30 | 10 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 1 | 0 | 6 | 1 | 8 | 2 | 1 | 0 | 0 | 0
INSOMNIA (Psychiatric disorders) | 3 | 0 | 0 | 6 | 0 | 10 | 2 | 0 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3 | 3 | 11 | 5 | 16 | 3 | 0 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 10 | 4 | 3 | 11 | 7 | 12 | 12 | 3 | 0 | 0 | 0
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 2 | 5 | 2 | 6 | 0 | 0 | 0 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 7 | 1 | 11 | 1 | 0 | 0 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 7 | 7 | 11 | 9 | 0 | 0 | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 9 | 11 | 6 | 13 | 14 | 15 | 19 | 6 | 0 | 0 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 4 | 0 | 7 | 7 | 1 | 8 | 3 | 8 | 2 | 1 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 3 | 3 | 0 | 8 | 8 | 9 | 9 | 0 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 9 | 0 | 3 | 16 | 11 | 21 | 15 | 3 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial